CLINICAL TRIAL: NCT00107289
Title: Open Access Protocol of Targeted Radiotherapy With I-metaiodobenzylguanidine (I-MIBG) in Patients With Resistant Neuroblastoma or Malignant Chromaffin Cell Tumors
Brief Title: Iodine I 131 Metaiodobenzylguanidine in Treating Patients With Recurrent, Progressive, or Refractory Neuroblastoma or Malignant Pheochromocytoma or Paraganglioma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-148; MSKCC-04148
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Neuroblastoma; Pheochromocytoma
Keywords: metastatic pheochromocytoma; recurrent pheochromocytoma; regional pheochromocytoma; recurrent neuroblastoma; 04-148
MeSH Terms: conditions — Neuroblastoma; Pheochromocytoma | interventions — 3-Iodobenzylguanidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Radiation (Experimental): Patients will be treated with IV 131I-MIBG using 1-2 high dose(s) or up to 16 low doses.
  Thyroid protection is commenced seven days (+/-2 days) prior to administration of 131I-MIBG and continued for up to 42 days after each 131I-MIBG treatment. Given that this is an open access protocol, re-enrollment is allowed per PI discretion. Patients who received this treatment previously are allowed to be re-enrolled if they meet the eligibility criteria. Re-enrollment can be to the same arm previously treated on (high dose versus low dose) or to the other arm. Patients will not be eligible for re-enrollment if they have already received 16 low doses or 4 high doses of 131I-MIBG.
  Interventions: Drug: iobenguane I 131

INTERVENTIONS:
Drug: iobenguane I 131 — A single dose of iodine I 131 metaiodobenzylguanidine (^131I-MIBG) IV over 30 minutes to 4 hours or for 15 minutes for smaller patients on day 0. Patients undergo radiation dosimetry following the first dose of ^131I-MIBG to determine if a second dose can be safely administered. Some patients may receive a second dose of iodine I 131 metaiodobenzylguanidine (^131I-MIBG) 6-8 weeks after the first dose. In some scenarios, extended time will be allowed before the second dose of 131I-MIBG for additional recovery and possible bridging therapy. If response is achieved and patients do not experience major toxicity. After blood radioactivity has fallen below 1 μCi/mL, patients may undergo autologous stem cell transplantation. After completion of study treatment, patients are followed at 4-6 weeks after ^131I-MIBG administration and then every 3 months for up to 1 year. Once patients are off treatment on this protocol, they will begin long term follow up through 5 years from enrollment.

SUMMARY:
The purpose of this research study is to find how active and safe 131 I-MIBG is in patients with resistant neuroblastoma, malignant pheochromocytoma and malignant paraganglioma.

ELIGIBILITY:
Inclusion criteria for NB:

* Patients must have the diagnosis of NB in accordance with the International Criteria, i.e., either histopathology (confirmed by the MSKCC Department of Pathology) or BM involvement plus elevated urinary catecholamines.
* Must have a history of tumor progression or recurrence or failure to achieve complete response with standard therapy.
* Patients must have MIBG-avid NB and evaluable disease on MIBG scan at time of enrollment on protocol
* Prior Therapy: At least 2 weeks should have elapsed since any biologic therapy. Three weeks should have elapsed since last dose of chemotherapy.
* Age >1 year
* Determination that radiation safety restrictions during therapy period can be implemented.
* Stem cells: Patients for high does must have an autologous hematopoietic stem cell product cryopreserved and available for re-infusion after MIBG treatment. Patients for low dose do not require cryopreserved autologous hematopoietic stem cell product available. The minimum dose for peripheral blood stem cells is 2 X106 CD34+ cells/kg.
* Minimum life expectancy of eight weeks
* Signed informed consent indicating awareness of the investigational nature of this program.

Inclusion criteria for malignant CCT:

* Patients must have the diagnosis of malignant CCT i.e. malignant pheochromocytoma or malignant paraganglioma
* Patients must have MIBG-avid malignant CCT and evaluable disease on MIBG scan at time of enrollment on protocol
* Prior Therapy: At least 2 weeks should have elapsed since any biologic therapy. Three weeks should have elapsed since last dose of chemotherapy.
* Age between 1 and 21 years and able to cooperate with radiation safety restrictions during therapy period
* Stem cells: Patients must have an autologous hematopoietic stem cell product cryopreserved and available for re-infusion after MIBG treatment. The minimum dose for peripheral blood stem cells is 2 X106 CD34+ cells/kg.
* Minimum life expectancy of eight weeks.
* Signed informed consent indicating awareness of the investigational nature of this program.

Exclusion Criteria:

* Severe major organ toxicity. Specifically, renal, cardiac, hepatic, pulmonary, gastrointestinal and neurologic toxicity should all be grade 2 or less. A grade 3 hearing deficit is acceptable.
* Active serious infections not controlled by antibiotics.
* Pregnant women are excluded for fear of danger to the fetus. Therefore negative pregnancy test is required for all women of child-bearing age, and appropriate contraception is used during the study period.
* Inability or unwillingness to comply with radiation safety procedures or protocol requirements.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Response (complete or partial) | 2 years

SECONDARY OUTCOMES:
Correlation between tumor self-absorbed dose and response and tumor volume decrease | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Basu, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Chu BP, Horan C, Basu E, Dauer L, Williamson M, Carrasquillo JA, Pandit-Taskar N, Modak S. Feasibility of Administering High-Dose (131) I-MIBG Therapy to Children with High-Risk Neuroblastoma Without Lead-Lined Rooms. Pediatr Blood Cancer. 2016 May;63(5):801-7. doi: 10.1002/pbc.25892. Epub 2016 Jan 15. PMID 26773712
- [Derived] Modak S, Zanzonico P, Carrasquillo JA, Kushner BH, Kramer K, Cheung NK, Larson SM, Pandit-Taskar N. Arsenic Trioxide as a Radiation Sensitizer for 131I-Metaiodobenzylguanidine Therapy: Results of a Phase II Study. J Nucl Med. 2016 Feb;57(2):231-7. doi: 10.2967/jnumed.115.161752. Epub 2016 Jan 7. PMID 26742708
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/